CLINICAL TRIAL: NCT02543489
Title: A Prospective, Post-market, Multi-center Comparative Study of the Efficacy of Flex Intramedullary(IM) Rod in Terms of Range of Motion (ROM) Improvement.
Brief Title: Flex Intramedullary Rod Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Stryker Japan K.K. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SJCR-OR-1103
Record Dates: First submitted 2015-08-10; First posted 2015-09-07 (Estimated); Last update posted 2018-09-14 (Actual); Status verified 2018-09

CONDITIONS: Osteoarthritis of the Knee; Arthroplasty, Replacement, Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Flex IM Rod (Other)
  Interventions: Device: Flex IM rod

INTERVENTIONS:
Device: Flex IM rod

SUMMARY:
The purpose of this study is to compare the effect of post-operative ROM between Flex IM rod and Rigid IM rod, to collect bone morphology of Japanese lower extremity and to research the incidence of overhung with Flex IM rod.

ELIGIBILITY:
Inclusion Criteria:

1. Patient has signed an Institutional Review Board (IRB) approved, study specific Informed Patient Consent Form.
2. Patient is a male or non-pregnant female age 20 years or older.
3. Patient is candidate for primary Total Knee Arthroplasty (TKA).
4. Patient whose preoperative range of motion (ROM) is over 110 degree.
5. Patient is willing and able to comply with postoperative scheduled clinical and radiographic evaluations and rehabilitation.

Exclusion Criteria:

1. Revision cases
2. Patients that use bone wedges or allograft due to bone loss.
3. Patient has a Body Mass Index (BMI) >40.
4. Patient has an active or suspected latent infection in or about the affected knee joint at time of study device implantation.
5. Patient has a neuromuscular or neurosensory deficiency, which limits the ability to evaluate the safety and efficacy of the device.
6. Patient is diagnosed with a systemic disease (e.g. Lupus Erythematosus) or a metabolic disorder (e.g. Paget's Disease) leading to progressive bone deterioration.
7. Patient is immunologically suppressed or receiving steroids in excess of normal physiological requirements (e.g. > 30 days).
8. Patient has failed unicondylar knee prosthesis.
9. Patient has a known sensitivity to device materials.
10. Patient who are inappropriate for participating in the study in the judgment of the investigator.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2012-12; Primary Completion 2019-09 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
Maximum postoperative flexion angle | 48 weeks after surgery

SECONDARY OUTCOMES:
Quality of life as assessed by36-Item Short-Form Health Survey (SF-36)questionnaire | 4 weeks , 24 weeks and 48 weeks after surgery
Japanese Knee Osteoarthritis Measure(JKOM) | 4 weeks , 24 weeks and 48 weeks after surgery
Knee Society Scale (KSS) | 4 weeks , 24 weeks and 48 weeks after surgery
Range of Motion (ROM) | 4 weeks , 24 weeks and 48 weeks after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Yasuyuki Inatsugu, Study Director — Stryker Japan
Locations (3):
- Japan (3):
  - Hyogo College of Medicine Hospital, Nishinomiya, Hyōgo
  - Saiseikai Yokohama East Hospital, Yokohama, Kanagawa
  - Osaka General Medical Center, Osaka